CLINICAL TRIAL: NCT06775483
Title: Evaluation of JSKN016 in the Treatment of Advanced Non-small Cell Lung Cance： a Phase II Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN016-201
Record Dates: First submitted 2024-12-30; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part I: Cohort 1（JSKN016） (Experimental): Enrolled subjects with harboring sensitive EGFR mutations who have already received tyrosine kinase inhibitor (TKI) therapy.Receive JSKN016 monotherapy , administered intravenously at the dosage specified in the protocol.
  Interventions: Drug: JSKN016
- Part I: Cohort 2（JSKN016） (Experimental): Enrolled subjects with negative driver genes who have already received immunotherapy. Receive JSKN016 monotherapy , administered intravenously at the dosage specified in the protocol.
  Interventions: Drug: JSKN016
- Part I: Cohort 3（JSKN016） (Experimental): Enrolled subjects with positive driver genes who have failed standard therapy.Receive JSKN016 monotherapy , administered intravenously at the dosage specified in the protocol.
  Interventions: Drug: JSKN016
- Part II：Cohort A（JSKN016） (Experimental): Receive JSKN016 monotherapy , administered intravenously at the dosage specified in the protocol.
  Interventions: Drug: JSKN016
- Part II：Cohort B（Docetaxel） (Active Comparator): Receive Docetaxel monotherapy , administered intravenously at the dosage specified in the protocol.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: JSKN016 — Administered intravenously according to protocol.
  Arms: Part I: Cohort 1（JSKN016）; Part I: Cohort 2（JSKN016）; Part I: Cohort 3（JSKN016）; Part II：Cohort A（JSKN016）
Drug: Docetaxel — Administered intravenously according to protocol.
  Arms: Part II：Cohort B（Docetaxel）

SUMMARY:
This is a Phase II clinical study conducted in China to evaluate the treatment of advanced non-small cell lung cancer with JSKN016. The enrolled subjects are all in the locally advanced or metastatic stage of non-small cell lung cancer.The study is divided into two parts. The main objective of part I is to assess the efficacy and safety of JSKN016 in selected subjects with advanced non-small cell lung cancer. The main objective of part II is to compare the efficacy of JSKN016 and docetaxel in subjects with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a Phase II clinical study conducted in China to evaluate the treatment of advanced non-small cell lung cancer with JSKN016. The enrolled subjects are all in the locally advanced or metastatic stage of non-small cell lung cancer.The study is divided into two parts. The main objective of part I is to assess the efficacy and safety of JSKN016 in selected subjects with advanced non-small cell lung cancer. The main objective of part II is to compare the efficacy of JSKN016 and docetaxel in subjects with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form.
2. Age ≥ 18 years old, male or female.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
4. Expected survival ≥ 3 months.
5. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) that is not suitable for radical surgery and/or radical radiotherapy, and meets one of the following conditions: EGFR sensitive mutations, and failed treatment with EGFR-TKI; Driver gene negative, treated with PD-1/L1 inhibitors and a platinum-containing chemotherapy and treatment failure; Positive driver gene, failure of corresponding standard therapy;
6. At least one extracranial measurable lesion at baseline according to RECIST 1.1 criteria.
7. Recently archived or fresh tumor tissue samples are available.
8. Have good organ function.
9. Have no current birth plans and agree to contraception during the trial.

Exclusion Criteria:

1. Presence of any small cell carcinoma component in histopathology.
2. Subjects with other malignant tumors within 5 years prior to enrollment, and other tumors have been cured through local therapy, such as cured cutaneous squamous cell carcinoma, basal cell carcinoma, non-primary invasive bladder cancer, and prostate/cervical/breast cancer in situ.
3. Presence of brainstem, meningeal metastases, spinal cord metastases or compression, leptomeningeal metastases, or history of carcinomatous meningitis; Presence of active brain metastases.
4. During the screening period, imaging shows that the tumor invades, compresses, or occurs in the surrounding important organs (such as the heart and pericardium, trachea, esophagus, superior vena cava, etc.) or there is a risk of esophageal tracheal fistula or esophageal pleural fistula.
5. Adequate washout of previous therapy before the first dose.
6. Gastrointestinal abnormalities with obvious clinical manifestations.
7. Presence of clinically severe respiratory impairment caused by pulmonary disease complications.
8. Presence of cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
9. Prior treatment with topoisomerase I inhibitors (e.g., irinotecan, topotecan), antibody-drug conjugates containing topoisomerase I inhibitors (e.g., DS-8201, HER3-DXd, DS-1062), or targeting TROP2 or HER3.
10. Previous treatment with docetaxel.
11. Have an uncontrolled infection, a history of immunodeficiency, a positive human immunodeficiency virus (HIV) test, or a history of AIDS.
12. Previous history of allogeneic bone marrow or organ transplantation.
13. Known allergy to any component of the study drug, and previous history of severe allergic reaction to other antibody drugs.
14. Pregnant and/or lactating females.
15. Have local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which can lead to higher medical risk and/or uncertainty in survival evaluation, such as tumor leukemia response , cachexia manifestations, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01-17 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by the investigator per RECIST v1.1 | Up to 24months
  Objective response rate (ORR) was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST v1.1）
Safety reflected by AE | Up to 24months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
DOR assessed by the investigator per RECIST v1.1 | Up to 24months
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR assessed by the investigator per RECIST v1.1 | Up to 24months
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR assessed by the investigator per RECIST v1.1 | Up to 24months
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
PFS assessed by investigator per RECIST v1.1 | Up to 24months
  Progression-free survival (PFS) is defined as the time from the date of initial administration till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).
OS | Up to 24months
  Overall Survival (OS) is defined as the time from the date of initial administration till death due to any cause.
Cmax of JSKN016 | Up to 24months
  Maximum (Peak) Observed blood Concentration (Cmax) of JSKN016 Following First Dose
AUC of JSKN016 | Up to 24months
  The blood PK parameters of JSKN016 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Tmax of JSKN016 | Up to 24months
  Time of Maximum blood Concentration (Tmax) of JSKN016 Following First Dose
ADA | Up to 24months
  Number of subjects with detectable anti-drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Overall Officials: Li zhang, Principal Investigator — Sun Yat-sen University